CLINICAL TRIAL: NCT00865124
Title: Role of Mineralocorticoid Receptor in Diabetic Cardiovascular Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Gail Kurr Adler, Associate Professor of Medicine, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2007-P-000564; 1R01HL087060-01A2 (NIH)
Record Dates: First submitted 2009-03-17; First posted 2009-03-19 (Estimated); Results first posted 2017-06-14 (Actual); Last update posted 2017-06-14 (Actual); Status verified 2017-05

CONDITIONS: Type 2 Diabetes Mellitus; Vascular Disease
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Vascular Diseases | interventions — Spironolactone; Hydrochlorothiazide; Potassium

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Spironolactone (mineralocorticoid receptor [MR] blockade) (Experimental)
  Interventions: Drug: Spironolactone
- Hydrochlorothiazide + potassium (Active Comparator)
  Interventions: Drug: Hydrochlorothiazide + potassium
- Placebo capsule (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Spironolactone — 25 mg capsule daily for 6 months
  Arms: Spironolactone (mineralocorticoid receptor [MR] blockade)
Drug: Hydrochlorothiazide + potassium — hydrochlorothiazide (HCTZ) + potassium, 12.5 mg/10 milliequivalents (mEq) capsule daily
  Arms: Hydrochlorothiazide + potassium
Other: Placebo — Placebo capsule daily
  Arms: Placebo capsule

SUMMARY:
Aldosterone is a significant mediator of cardiovascular injury associated with heart failure and the cardiovascular benefits of mineralocorticoid receptor blockade are additive to those of angiotensin converting enzyme inhibitors or angiotensin II (ANGII) receptor blockers. This study will test the hypothesis that mineralocorticoid receptor (MR) antagonists exert beneficial cardiovascular effects, specifically by decreasing vascular injury and improving vascular function. A randomized, double-blind study will be conducted, in which participants with Type 2 Diabetes Mellitus will undergo a series of assessments to test heart, blood vessel, and kidney function at baseline, and after 2 and 6 months of treatment with one of the following drugs:

1. spironolactone
2. hydrochlorothiazide (HCTZ) plus potassium
3. placebo

In the event of insufficient funds, randomization to the placebo arm will be stopped and primary assessment of outcomes will occur at baseline and after 6 months of treatment.

ELIGIBILITY:
Inclusion Criteria:

* age 18-70 years
* type 2 diabetes mellitus
* with or without hypertension

Exclusion Criteria:

* ischemic changes on resting electrocardiogram,
* clinical evidence of heart disease (angina, heart failure, unstable angina),cerebrovascular or peripheral vascular disease,
* significant cardiac arrhythmias,
* aortic stenosis,
* 2nd or 3rd degree atrio-ventricular block, sinus node disease, or symptomatic bradycardia,
* bronchospastic lung disease with active wheezing,
* known hypersensitivity to adenosine,
* hemoglobin A1C (HbA1c) > 8.5%, *
* gout (If not already taking HCTZ),
* the use of Rosiglitazone,**
* estimated glomerular filtration rate (eGFR) < 60 ml/min,
* serum potassium > 5.0 mmol/L,
* use of potassium-sparing diuretics,**
* current smoker,*
* pregnancy,
* renal disease not related to diabetes mellitus,
* uncontrolled hypertension, systolic blood pressure (BP) >160 mm Hg and diastolic BP >100 mm Hg,*
* use of cyclic hormone replacement therapy
* past intolerance of angiotensin-converting enzyme (ACE) inhibitor therapy
* other major medical illnesses. Participants with evidence of a previous myocardial infarction on the first adenosine-stimulated positron emission tomography (PET) study will be withdrawn from the study.
* Screening systolic blood pressure < 105 mm Hg off of anti-hypertensive medications

  * Participants can enroll in study and proceed with in-patient evaluations if during the run-in period adjustments of medications, diet and habits lead to improved glucose control [equivalent to HbA1c <8.5%, controlled hypertension and cessation of smoking.

    * Participants who are currently taking these medications will not qualify for a screening visit. If medications were recently stopped by the participant's physician, he or she may be screened but the baseline assessment protocol must occur 3 months after stopping.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2008-09; Primary Completion 2013-08 (Actual); Study Completion 2014-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gail K Adler, MD, PhD, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Haas AV, Rosner BA, Kwong RY, Rao AD, Garg R, Di Carli MF, Adler GK. Sex Differences in Coronary Microvascular Function in Individuals With Type 2 Diabetes. Diabetes. 2019 Mar;68(3):631-636. doi: 10.2337/db18-0650. Epub 2018 Nov 8. PMID 30409780
- [Derived] Garg R, Rao AD, Baimas-George M, Hurwitz S, Foster C, Shah RV, Jerosch-Herold M, Kwong RY, Di Carli MF, Adler GK. Mineralocorticoid receptor blockade improves coronary microvascular function in individuals with type 2 diabetes. Diabetes. 2015 Jan;64(1):236-42. doi: 10.2337/db14-0670. Epub 2014 Aug 14. PMID 25125488

RESULTS

PARTICIPANT FLOW:
Groups:
- Spironolactone (MR Blockade): 25 mg capsule daily for 6 months
Period: Overall Study
Arm/Group | Spironolactone (MR Blockade) | Hydrochlorothiazide + Potassium | Placebo
Started | 27 | 25 | 17
Completed | 23 | 24 | 17
Not Completed | 4 | 1 | 0
Not completed — Physician Decision | 2 | 1 | 0
Not completed — Withdrawn consent | 2 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All participants who completed the study.
Groups:
- Spironolactone (MR Blockade): Spironolactone: 25 mg capsule daily for 6 months
- Hydrochlorothiazide + Potassium: Hydrochlorothiazide + potassium: hydrochlorothiazide (HCTZ) + potassium, 12.5 mg/10 mEq capsule daily
- Total: Total of all reporting groups
Arm/Group | Spironolactone (MR Blockade) | Hydrochlorothiazide + Potassium | Placebo Capsule | Total
Number analyzed (Participants) | 23 | 24 | 17 | 64
Age, Continuous [Mean (Standard Deviation); unit: years] | 56 (6) | 53 (7) | 55 (10) | 54.72 (7.66)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 11 | 7 | 24
  Male | 17 | 13 | 10 | 40

OUTCOME MEASURES:

1. Primary Outcome: Change in Coronary Flow Reserve From Baseline to 6 Months
Description: Coronary flow reserve (CFR), or myocardial perfusion reserve, was assessed via cardiac positron emission tomography (PET). CFR is the ratio of adenosine-stimulated blood flow through myocardium to resting blood flow through myocardium. An improvement in coronary flow reserve is beneficial.
Time Frame: Baseline and six months
Population: All participants with data available for this outcome measure.
Measure: Mean (Standard Deviation); unit: ratio
Groups:
- Hydrochlorothiazide + Potassium: Hydrochlorothiazide (HCTZ) + potassium, 12.5 mg/10 mEq capsule daily
Arm/Group | Spironolactone (MR Blockade) | Hydrochlorothiazide + Potassium | Placebo
Number analyzed (Participants) | 22 | 22 | 16
ratio | 0.33 (0.83) | -0.10 (0.65) | 0.02 (1.03)

2. Secondary Outcome: Change in Mitral Annulus Velocities on Tissue Doppler (Delta E/e' Ratio), a Measure of Diastolic Function
Description: Diastolic function was assessed via tissue doppler imaging (TDI) by echocardiography to determine left ventricular diastolic function before and after 6 months of treatment.
Time Frame: Baseline and six months
Population: All participants with data available for this outcome measure.
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Spironolactone (MR Blockade) | Hydrochlorothiazide + Potassium | Placebo
Number analyzed (Participants) | 23 | 24 | 17
ratio | 0.02 (1.61) | 0.06 (1.35) | 0.64 (1.95)

3. Secondary Outcome: Mitral Annulus Velocities on Tissue Doppler (Delta E/e' Ratio), a Measure of Diastolic Function (With Angiotensin II)
Description: Diastolic function was assessed via tissue doppler imaging (TDI) by echocardiography to determine left ventricular diastolic function before and after 6 months of treatment; and in response to acute administration (3 nanograms/kg/min for 60 min) of the vasoactive agent, Angiotensin II.
Time Frame: Baseline and six months
Population: All participants with data available for this outcome measure at the given time-point.
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Spironolactone (MR Blockade) | Hydrochlorothiazide + Potassium | Placebo
Number analyzed (Participants) | 27 | 25 | 17
ratio
  Pre-treatment, E/e', baseline: number analyzed (Participants) | 26 | 23 | 15
  Pre-treatment, E/e', baseline | 6.67 (1.93) | 6.72 (1.93) | 6.55 (2.24)
  Pre-treatment, E/e', Post-ANGII: number analyzed (Participants) | 24 | 17 | 12
  Pre-treatment, E/e', Post-ANGII | 7.09 (1.96) | 7.06 (1.66) | 6.70 (3.08)
  6 months post-treatment, E/e', baseline: number analyzed (Participants) | 22 | 21 | 15
  6 months post-treatment, E/e', baseline | 6.76 (1.57) | 7.03 (1.83) | 7.35 (2.26)
  6 months post-treatment, E/e', Post-ANGII: number analyzed (Participants) | 17 | 15 | 12
  6 months post-treatment, E/e', Post-ANGII | 6.28 (2.53) | 5.83 (2.82) | 7.48 (1.59)

4. Secondary Outcome: Change in Renal Plasma Flow
Description: Renal vasculature was assessed by examining renal plasma flow, or para-aminohippurate (PAH) clearance, basally and in response to acute administration (3 nanograms/kg/min for 60 min) of the vasoactive agent, Angiotensin II.
Time Frame: Baseline and six months
Population: All participants with data available for this outcome measure at the given time-point.
Measure: Mean (Standard Deviation); unit: mL/min/1.73m^2
Arm/Group | Spironolactone (MR Blockade) | Hydrochlorothiazide + Potassium | Placebo
Number analyzed (Participants) | 27 | 25 | 17
mL/min/1.73m^2
  Pre-treatment, PAH clearance, baseline: number analyzed (Participants) | 26 | 23 | 17
  Pre-treatment, PAH clearance, baseline | 527 (76) | 508 (82) | 518 (108)
  Pre-treatment, PAH clearance, Post-ANGII: number analyzed (Participants) | 24 | 18 | 14
  Pre-treatment, PAH clearance, Post-ANGII | 442 (75) | 417 (49) | 436 (97)
  6 months post-treatment, PAH clearance, baseline: number analyzed (Participants) | 21 | 22 | 17
  6 months post-treatment, PAH clearance, baseline | 518 (97) | 500 (80) | 491 (87)
  6 months post-treatment, PAH clearance, Post-ANGII: number analyzed (Participants) | 18 | 17 | 13
  6 months post-treatment, PAH clearance, Post-ANGII | 423 (89) | 415 (61) | 427 (99)

ADVERSE EVENTS:
Time Frame: 6 months
Description: Adverse events are reported for participants who received study treatment.
Arm/Group | Spironolactone (MR Blockade) | Hydrochlorothiazide + Potassium | Placebo
All-Cause Mortality (participants affected / at risk) | 0/27 | 0/25 | 0/17
Serious Adverse Events (participants affected / at risk) | 2/27 | 0/25 | 0/17
Other Adverse Events (participants affected / at risk) | 6/27 | 5/25 | 3/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Spironolactone (MR Blockade) (N=27) | Hydrochlorothiazide + Potassium (N=25) | Placebo (N=17)
Pulmonary embolism (Vascular disorders) | 1 | 0 | 0
Increased potassium (Investigations) | 1 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Spironolactone (MR Blockade) (N=27) | Hydrochlorothiazide + Potassium (N=25) | Placebo (N=17)
Vomiting (Gastrointestinal disorders) | 0 | 1 | 0
Reversible ischemia (Cardiac disorders) | 1 | 0 | 2
Hyperglycemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Injection site reaction (Injury, poisoning and procedural complications) | 1 | 0 | 0
Dilated pulmonary artery (Vascular disorders) | 1 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 1 | 0
Stomach pain (Gastrointestinal disorders) | 0 | 1 | 0
Lung nodule (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0
Renal cyst (Renal and urinary disorders) | 0 | 0 | 1
Liver lesion (Hepatobiliary disorders) | 0 | 0 | 1
Thoracic vertebral hemangioma (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Nodular opacity in the lung (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pericardial effusion (Cardiac disorders) | 1 | 0 | 0
Stress-induced ischemia (Cardiac disorders) | 0 | 2 | 0
Vertebral degeneration (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Atrial septal aneurysm (Cardiac disorders) | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes